CLINICAL TRIAL: NCT00186732
Title: Pfannenstiel Incision Closure: Subcuticular Suture Versus Surgical Staples
Brief Title: Comparison of Subcuticular Suture Versus Surgical Staples for Closure of Pfannenstiel Skin Incisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-2484
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Pain, Postoperative; Gynecologic Surgical Procedures; Obstetric Surgical Procedures
Keywords: wound closure; Pfannenstiel incision; surgical staples; subcuticular suture
MeSH Terms: conditions — Pain, Postoperative | interventions — Sutures

INTERVENTIONS:
Procedure: Subcuticular Suture
Procedure: Surgical Staples

SUMMARY:
This study compares methods of closure for Pfannenstiel incisions commonly used during gynecological and obstetrical surgery. Patients are assigned to closure by either surgical staples or a buried suture. Information is collected on the day of surgery, post-operative day two and at the six-week follow up visit. The amount of pain and cosmetic result are compared. Infection rates will also be monitored for the two groups.

The study hypothesis is as follows: subcuticular (buried) sutures as compared to surgical staples lead to decreased post-operative pain and improved cosmetic result. Infection rates are similar for both groups.

DETAILED DESCRIPTION:
There is little evidence in the literature to guide the choice of closure material for Pfannenstiel laparotomy. Currently this decision is based primarily on physician preference. Physicians differ greatly in their view on which is better. This is based on personal habit and experience and not on scientific evidence. Specifically in the field of obstetrics and gynecology there has only been one randomized trial of approximately 60 patients undergoing cesarean section comparing subcuticular suture vs surgical staples for closure of their Pfannenstiel skin incisions (Frishman et al., 1997). This study showed that Pfannenstiel skin incisions closed with subcuticular closure following cesarean section result in less postoperative pain and are more cosmetically appealing as compared to incisions closed with staples.

This randomized controlled study will compare closure of Pfannenstiel incisions using either subcuticular absorbable suture or surgical staples. It will examine two separate populations - those undergoing cesarean section and those undergoing gynecological surgery such as hysterectomy. These patient groups will be analyzed separately as their demographic characteristics tend to be quite different. The primary outcome will be postoperative pain. Cosmetic result will be a secondary outcome. Cosmesis will be rated both by the patient and the physician. Infection rates are also of great interest although it is unlikely that this study will achieve adequate power to show a statistically significant difference in results. Other outcomes of interest include overall patient satisfaction, total operating room time and length of hospital stay. Patient's body mass index will also be recorded and analyzed to determine whether it affects results in both intervention groups.

There will be a minimum of 144 patients total in the cesarean section group and 144 patients total in the gynecological surgery group - 72 randomized to staples and 72 randomized to subcuticular suture for each group. Thus the entire study will involve approximately 288 patients.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing gynecological or obstetrical surgery
* Pfannenstiel skin incision

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2005-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Pain

SECONDARY OUTCOMES:
Cosmesis
Infection rates
Length of stay OR time
Overall patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Cara A Donnery, MD, Principal Investigator — McMaster University Obstetrics and Gynecology Resident; Richard Persadie, MD, Principal Investigator — Staff Doctor: St. Joseph's Healthcare, Hamilton
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada